CLINICAL TRIAL: NCT02455453
Title: Assessment of Functional Status of Estrogen Receptors in Breast Cancer by Positron Emission Tomography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201411005; 5R01CA195450-03 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic FFNP-PET/CT Scan (Experimental): * (2) 18F-FFNP-PET/CT scans
    * First one prior to estradiol challenge test
    * Second one immediately following one day of estradiol challenge test
  * (1) FDG-PET/CT scan at screening
  * The estradiol challenge test will consist of administering a total of 6 mg of estradiol dosed orally as three 2 mg tablets with each tablet being administered approximately 8 hours apart and within a 24 hour period. This estradiol medication will be provided to the patient by the study.
  Interventions: Drug: 18F-FFNP; Device: CTI/Siemens Biograph 40 PET/CT Scanner; Drug: Estradiol; Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FFNP
  Other Names: 21-18F-fluoro-16α,17α-[(R)-(1'-α-furylmethylidene)dioxy]-19-norpregn-4-ene-3,20-dione
Device: CTI/Siemens Biograph 40 PET/CT Scanner — * Will include (1) 18-FDG-PET/CT scan
  * Will include (2) 18F-FFNP-PET/CT scans
Drug: Estradiol
Drug: 18F-FDG

SUMMARY:
The purpose of this study is to evaluate the uptake of a radioactive tracer 21-18F-fluoro-16α,17α-[(R)-(1'-α-furylmethylidene)dioxy]-19-norpregn-4-ene-3,20-dione (FFNP) uptake, which binds to breast cancer progesterone receptors (PgRs) on a PET/CT scan before and after administration of estradiol for one day (estrogen challenge) to determine if the change in uptake is a predictor of response to endocrine therapy (ET) in patients with hormone-sensitive estrogen receptor positive (ER+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer. Estradiol is the most potent of the naturally occurring estrogens, and can be administered to treat menopausal symptoms and also sometimes to treat metastatic breast cancer. The investigators propose to study patients with biopsy-proven newly diagnosed, locally advanced, metastatic, or recurrent breast cancer who are going to be treated with endocrine therapy (ET) (tamoxifen,aromatase inhibitors or fulvestrant as standard of care therapy.

Subjects will undergo a total of two FFNP-PET/CT scans; one before and a second one immediately following the one day estradiol challenge before the start of standard of care ET. The estradiol challenge will consist of administering a total of 6 mg of estradiol orally (three doses of 2 mg each) given at approximately 8 hour intervals and over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be postmenopausal defined as meeting one or more of the following:

  * Age ≥ 60 years
  * Amenorrheic for at least 12 months
  * Surgically sterile- having undergone bilateral oophorectomy,
  * FSH level in postmenopausal range according to institutional standards (note follicle-stimulating hormone (FSH) laboratory testing must be ordered as standard of care to determine optimal treatment and should not be ordered simply to confirm eligibility to this study)
  * OR Pre-menopausal for whom standard estradiol treatment (ET) is planned with ovarian suppression (imaging on study should be completed prior to start of ovarian suppression)
* Patient must have histological or cytological confirmed breast cancer and fall into one of the following categories:

  * New diagnosis with plans for at least 6 months of neoadjuvant ET or any amount of neoadjuvant ET if surgery is planned as this will be used for response assessment .
  * Patients with newly diagnosed metastatic breast cancer or patient with known metastatic disease who has progressed while on therapy (no washout period is needed if the patient was treated with AIs or chemotherapy, but 2 months washout period is needed if the patient was treated with tamoxifen) who are going to be treated with ET.
* Patient must have any one of the following types of breast cancer (primary or metastatic): ER+/PgR+/HER2- or ER+/PgR-/HER2-.

  * ER+ is defined as Allred score of at least 4 and greater.
  * PgR+ is defined as Allred score of at least 4 and greater.
  * Immunohistochemistry (IHC) is the primary assay methodology for HER2. HER2- refers to HER2 of 0, 1+ by IHC or negative by fluorescence in situ hybridization (FISH)
* Patient must have at least one measurable lesion according to RECIST 1.1 by radiological evaluation (ultrasound, mammography, MRI, CT, PET) or physical examination.

  * Patients with evaluable osseous metastasis that are lytic or mixed lytic-sclerotic are eligible.
  * Patients with hepatic lesions may be eligible provided the location of the lesion is peripheral or not too close to hepatic ducts. Decision on hepatic lesion eligibility will be made by the principal investigator or sub-investigator after careful review of all available imaging to ensure evaluation of the lesion will not be obscured by normal hepatobiliary excretion of 18F-FFNP.
* Patient must be able to understand and willing to sign a written informed consent document.
* Prior chemotherapy or endocrine therapy is allowed
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or, based on the judgment of the treating medical oncologist, can tolerate imaging and at least 6 months of ET
* The patient should have a life expectancy of > 6 months.

Exclusion Criteria:

* Patient with other invasive malignancies, with the exception of non-melanoma skin cancer or cervical carcinoma in-situ, who had (or have) any evidence of the other cancer present within the last 5 years
* Unable to tolerate up to 60 min of PET imaging per imaging session.
* Patients with non-measurable non-evaluable lesions such as pleural effusion are not eligible to participate.
* Patients with vertebral lesions that, in the opinion of the Principal Investigator and the treating medical oncologist, pose an imminent risk for cord compression.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dehdashti F, Wu N, Ma CX, Naughton MJ, Katzenellenbogen JA, Siegel BA. Association of PET-based estradiol-challenge test for breast cancer progesterone receptors with response to endocrine therapy. Nat Commun. 2021 Feb 2;12(1):733. doi: 10.1038/s41467-020-20814-9. PMID 33531464
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic FFNP-PET/CT Scan
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic FFNP-PET/CT Scan
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 60.0 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Primary Tumor FFNP Uptake Before and After Estradiol Challenge as Measured by Percent Change in Standardized Uptake Value (SUV)
Time Frame: Completion of second FFNP-PET/CT scan (up to 4 weeks)
Population: 2 participants were not included in this outcome measure as the liver background was too high in both participants.
Measure: Median (Full Range); unit: percent change in SUV
Arm/Group | Diagnostic FFNP-PET/CT Scan
Number analyzed (Participants) | 45
percent change in SUV | 11.0 [-46.0 to 306.0]

2. Primary Outcome: Change in Secondary Tumor FFNP Uptake Before and After Estradiol Challenge as Measured by Percent Change in Standardized Uptake Value (SUV)
Time Frame: Completion of second FFNP-PET/CT scan (up to 4 weeks)
Population: 12 participants were not included in this outcome measure as they did not have a secondary tumor location and 2 participants were not included in this outcome measure as the liver background was too high in both participants.
Measure: Median (Full Range); unit: percent change in SUV
Arm/Group | Diagnostic FFNP-PET/CT Scan
Number analyzed (Participants) | 33
percent change in SUV | 15.0 [-48.0 to 306.0]

3. Secondary Outcome: Heterogeneity of Tumor FFNP Uptake as Measured by Number of Participants With Heterogenous Response
Description: As measured visually in known lesion by recording presence or absence of uptake with note of any changes between scans
Time Frame: Completion of second FFNP-PET/CT scan (up to 4 weeks)
Population: 2 participants were not included in this outcome measure as the liver background was too high in both participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic FFNP-PET/CT Scan
Number analyzed (Participants) | 45
Participants | 6

ADVERSE EVENTS:
Time Frame: For FFNP-PET/CT imagings, participants were contacted by phone or in person approximately 24 +/- 6 hours after the injection of 18FFNP to assess for adverse events as related to 18F-FFNP injection, or PET/CT imaging. Any adverse events that occurred within 24 hours of administration of 18F-FFNP or within 24 hours of the first dose of estradiol which are graded related or possibly related were reported.
Arm/Group | Diagnostic FFNP-PET/CT Scan
All-Cause Mortality (participants affected / at risk) | 5/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 11/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic FFNP-PET/CT Scan (N=47)
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Oral dysesthesia (Gastrointestinal disorders) | 1
Abdominal cramping (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Shoulder/joint pain (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 2
Bug bite or welt (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT02455453/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02455453/ICF_001.pdf